CLINICAL TRIAL: NCT03820895
Title: Assessment of Serum Vitamin D Levels in Surgical Adolescent Idiopathic Scoliosis Patients
Brief Title: Vitamin D Levels in Adolescent Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Security Forces Hospital (Other)
Collaborators: King Saud University (Other)
Responsible Party: Principal Investigator, Raheef Alatassi, Orthopedic Surgeon, Security Forces Hospital
Other Study IDs: vit d in AIS
Record Dates: First submitted 2019-01-26; First posted 2019-01-29 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Scoliosis Idiopathic; Vitamin D Deficiency; BMD
Keywords: vitamin D; Cobb angle; alkaline phosphatase
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Hematologic Tests; X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood test — Serum 25-hydroxyvitamin D 25(OH) D levels were measured for Vitamin D status, by electrochemiluminescence immunoassay (Roche, USA). Cobb's angle measurement was done by measuring the major spinal curve and was taken from the upper end vertebra to the lower end vertebra through an x-ray for all the patients included in the study.
  Other Names: X-ray

SUMMARY:
This study aims to estimate the prevalence of vitamin D insufficiency among patients with adolescent idiopathic scoliosis, to calculate the differences in serum vitamin D levels, Cobb angles, spinal bone mass densities, and serum alkaline phosphatase levels between genders in the sample, and to assess the possibility of a correlation between any of these factors in those surgical patients.

DETAILED DESCRIPTION:
Adolescent Idiopathic Scoliosis (AIS) is a major public health problem and despite its relative rareness, it reduces the quality of life. It is three-dimensional deformity where there is a lateral curving of the spine. The prevalence rate is 0.47-5.2%. The degree of the spinal curvature is evaluated by the Cobb angle. A Cobb angle of more than 10-15° is considered pathological. AIS occurs mostly in adolescents between 10 and 25 years of age, and is more prevalent among females.

Scoliosis is considered severe and requires surgical intervention when the Cobb angle exceeds 40o.

The etiology of AIS is still unknown. Genetic and non-genetic factors have been attributed to cause AIS. Among non-genetic factors is bone mineral density (BMD), as bone quality plays an important role in the derangement of bony mechanical stability. The prevalence of AIS with osteoporosis is approximately 20-38%. Osteoporosis is known to lower the bone strength.

Vitamin D plays an essential role in maintaining a healthy mineralized skeleton. It helps with calcium absorption, and patients with a deficiency of Vitamin D can have difficulties in producing new bone and maintaining their bone strength.

In this study, the prevalence of vitamin D insufficiency among patients with AIS was evaluated. Gender differences in serum vitamin D levels, Cobb angles, BMD, and serum alkaline phosphatase levels were measured. Further correlation of Vitamin D with Cobb angles, BMD, and serum ALP levels was also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* AIS patients of either gender
* Aged between 10-25 years old
* Had Cobb angles of 40o or more (i.e. requiring corrective surgery)
* Had their serum vitamin D levels measured prior to their corrective surgery.

Exclusion Criteria:

* Patients with non-idiopathic scoliosis (such as congenital or neuromuscular condition)
* Younger than 10 years
* Older than 25 years of age
* Who did not have their serum vitamin D levels present on the system.

Ages: 10 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patient who suffer from AIS and are eligible for corrective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
measure vitamin D level in AIS patients | Baseline
  Serum 25-hydroxyvitamin D 25(OH) D levels were measured for Vitamin D status, by electrochemiluminescence immunoassay (Roche, USA).

SECONDARY OUTCOMES:
calculate Cobb's angle in AIS patients | Baseline
  done by measuring the major spinal curve and was taken from the upper end vertebra to the lower end vertebra through an x-ray for all the patients included in the study.
measure BMD values in AIS patients | Baseline
  were taken from the spine only by the use of a dual energy x-ray absorptiometry (DXA) scanner (Lunar, General Electric (GE) medical systems, UK)
measure Serum alkaline phosphatase (ALK) in AIS patients | Baseline
  measured using a biochemical auto-analyzer (Siemens health diagnostics, USA).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nowak R, Szota J, Mazurek U. Vitamin D receptor gene (VDR) transcripts in bone, cartilage, muscles and blood and microarray analysis of vitamin D responsive genes expression in paravertebral muscles of juvenile and adolescent idiopathic scoliosis patients. BMC Musculoskelet Disord. 2012 Dec 23;13:259. doi: 10.1186/1471-2474-13-259. PMID 23259508
- [Result] Gozdzialska A, Jaskiewicz J, Knapik-Czajka M, Drag J, Gawlik M, Ciesla M, Kulis A, Zarzycki D, Lipik E. Association of Calcium and Phosphate Balance, Vitamin D, PTH, and Calcitonin in Patients With Adolescent Idiopathic Scoliosis. Spine (Phila Pa 1976). 2016 Apr;41(8):693-7. doi: 10.1097/BRS.0000000000001286. PMID 27064335
- [Result] Konieczny MR, Senyurt H, Krauspe R. Epidemiology of adolescent idiopathic scoliosis. J Child Orthop. 2013 Feb;7(1):3-9. doi: 10.1007/s11832-012-0457-4. Epub 2012 Dec 11. PMID 24432052
- [Result] Al-Arjani AM, Al-Sebai MW, Al-Khawashki HM, Saadeddin MF. Epidemiological patterns of scoliosis in a spinal center in Saudi Arabia. Saudi Med J. 2000 Jun;21(6):554-7. PMID 11500705
- [Result] Yaman O, Dalbayrak S. Idiopathic scoliosis. Turk Neurosurg. 2014;24(5):646-57. doi: 10.5137/1019-5149.JTN.8838-13.0. PMID 25269032
- [Result] Adobor RD, Joranger P, Steen H, Navrud S, Brox JI. A health economic evaluation of screening and treatment in patients with adolescent idiopathic scoliosis. Scoliosis. 2014 Dec 6;9(1):21. doi: 10.1186/s13013-014-0021-8. eCollection 2014. PMID 25601889
- [Result] Lee WT, Cheung CS, Tse YK, Guo X, Qin L, Lam TP, Ng BK, Cheng JC. Association of osteopenia with curve severity in adolescent idiopathic scoliosis: a study of 919 girls. Osteoporos Int. 2005 Dec;16(12):1924-32. doi: 10.1007/s00198-005-1964-7. Epub 2005 Sep 15. PMID 16163440
- [Result] Al-Othman A, Al-Musharaf S, Al-Daghri NM, Krishnaswamy S, Yusuf DS, Alkharfy KM, Al-Saleh Y, Al-Attas OS, Alokail MS, Moharram O, Sabico S, Chrousos GP. Effect of physical activity and sun exposure on vitamin D status of Saudi children and adolescents. BMC Pediatr. 2012 Jul 3;12:92. doi: 10.1186/1471-2431-12-92. PMID 22759399
- [Derived] Alsiddiky A, Alfadhil R, Al-Aqel M, Ababtain N, Almajed N, Bakarman K, Awwad W, Alatassi R. Assessment of serum vitamin D levels in surgical adolescent idiopathic scoliosis patients. BMC Pediatr. 2020 May 11;20(1):202. doi: 10.1186/s12887-020-02114-9. PMID 32393207